CLINICAL TRIAL: NCT00481052
Title: The Protein Tyrosine Kinase Inhibitor Nilotinib as First-line Treatment of Ph+ Chronic Myeloid Leucemia (CML) in Early Chronic Phase: a Phase II Exploratory, Multicenter Study. GIMEMA Protocol CML 0307. EUDRACT 2007-000597-22.
Brief Title: Nilotinib as First-line Treatment of Ph+ CML in Early Chronic Phase
Acronym: CML0307
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML0307
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Adult; CML; Philadelphia positive; Nilotinib; early chronic phase; untreated or treated only with Hydroxyurea or Anagrelide; Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nilotinib

SUMMARY:
Treating Ph pos CML with Imatinib is very effective since the majority of the patients achieve a complete cytogenetic response and a major molecular response and are alive and progression-free after 5 years. However, the great majority of responding patients are not leukemia-free and may be at risk of progression, molecular, cytogenetic and clinical, at any time. In case of disease progression due to Imatinib failure, nilotinib has been found to be very effective, as expected from the preclinical profile of the drug, that is much more potent against BCR-ABL and inhibits nearly all the imatinib-resistant BCR-ABL mutants. For these reasons, nilotinib is going to be registered for the treatment of imatinib-resistant CMl patients. For the same reasons, nilotinib is expected to be more efficient than imatinib also front-line, based on the principle that we should aim at preventing the emergence of resistance better that at treating resistance once it has emerged. This expectation can be tested safely, because the "toxicity profile" of Nilotinib may be even more convenient than that of Imatinib, due to the lower frequency of edema and fluid retention.

DETAILED DESCRIPTION:
Study Phase:

Phase II, Prospective, multicentric, non randomized, open label

Objectives:

The primary objective of the trial is to investigate the cytogenetic and molecular effects of the protein tyrosine kinase (PTK) inhibitor nilotinib in the treatment of early chronic phase Ph+ CML.

The secondary objectives are:

To investigate in early CP Ph+ CML patients treated with nilotinib the clinical and the hematologic effects, the effect on bcr/abl point mutations, the kinetic of the response, the toxicity, the compliance to treatment and the dose density.

Study design:

This study is an open-label, multicenter, exploratory, Phase II study of nilotinib administered orally twice daily for one year. For the patients who will benefit an extension to 4 years is planned.

Visit Schedule and Assessments:

A visit with blood counts and differential and serum chemistry is due baseline, every 15 days for 3 months, hence every 30 days.

An ECG is due baseline, after 15 and 30 days, hence at 60, 90, 150, 240 and 360 days.

An echocardiogram is due baseline and at end-of-study (360 days) or early withdrawal.

A bone marrow aspirate is due baseline (cytology, cytogenetics and quantitative molecular biology), after 3 and 6 months (cytology and cytogenetics) and after 12 months (cytology, cytogenetics, quantitative molecular biology and mutational analysis).

A peripheral blood sample is due baseline, at 30, 60, 90, 180, 270 and 360 days for quantitative molecular biology.

After the end of the study (i.e. after one year) clinical, cytogenetic and molecular data are due every 6 months.

Biologic Monitoring:

Bone marrow and peripheral blood cells will be collected before, during and at the end of the study, stored at the central lab in Bologna and used for molecular assays that are listed in details in the protocol, with the exclusion of any test allowing the identification of patients genotype. The samples are kept for a minimum of 10 years and can be destroyed upon patient request. A specific consent form to the sample storage will be submitted to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cytologic and cytogenetic confirmed diagnosis of Ph+ CML.
* Age ≥ 18 years old
* Early CP (within 6 months from diagnosis)
* No prior treatment with any antileukemic drugs with the exception of Hydroxyurea (HU) and Anagrelide.
* WHO performance status of ≤ 2
* Normal serum level of potassium, total calcium corrected for serum albumin, magnesium and phosphorus, or correctable with supplements
* ALT and AST ≤ 2.5 x ULN or ≤ 5.0 x ULN if considered due to leukaemia.
* Alkaline phosphatase ≤ 2.5 x ULN unless considered due to leukemia.
* Serum bilirubin ≤ 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN
* Serum amylase ≤ 1.5 x ULN and serum lipase ≤ 1.5 x ULN.
* Written informed consent prior to any study procedures being performed.

Exclusion criteria:

* Impaired cardiac function, including LVEF < 45% as determined by MUGA scan or echocardiogram, uncontrolled congestive heart failure, uncontrolled hypertension
* History of myocardial infarction within three months, or uncontrolled angina pectoris.
* Significant electric heart abnormalities, including history or presence of significant ventricular or atrial tachyarrhythmias, congenital long QT syndrome and/or QTc > 450 msec on screening ECG (using the QTcF formula).
* Patients with ventricular pacemakers and clinically significant bradycardias.
* Patients with heart blocks.
* History of acute or chronic pancreatitis.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of nilotinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Use of therapeutic coumarin derivates (i.e. warfarin, acenocoumarol, phenprocoumon).
* Acute or chronic liver or renal disease considered unrelated to leukaemia
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes, active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
* Patients who are currently receiving treatment with any of the medications listed in Appendix E and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug. The medications listed in Appendix E have the potential to prolong QT, with the exception of HU and Anagrelide.
* Patients who have received any antileukemic agents and treatments, including HSCT, with the exception of HU and Anagrelide.
* Patients who have received any investigational drug ≤ 4 weeks.
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control. (Women of childbearing potential must have a negative serum pregnancy test within 48 hrs prior to administration of nilotinib). Post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
* Treatment with any hematopoietic colony-stimulating growth factors (e.g. G-CSF, GM-CSF) 1 week prior to starting study drug.
* Patients who have received immunotherapy 1 week prior to starting study drug or who have not recovered from side effects of such therapy.
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory).
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention.
* Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-06-23 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Complete cytogenetic response (CCgR ) rate | At 1 year

SECONDARY OUTCOMES:
The complete and the partial cytogenetic response rate | At 6 months
The major molecular response (MMR) rate | At 1 year
The kinetics of haematologic, cytogenetic and molecular response to AMN107 | At 1 year
The development of bcr-abl mutation during the treatment with AMN107 (number and type) | At 1 year
The safety and tolerability of nilotinib treatment at the dose of 300 mg b.i.d | At 1 year
To describe any SAE | At 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michele BACCARANI, Principal Investigator — Azienda Ospedaliera Universitaria -Policlincio S. Orsola-Malpighi
Locations (22):
- Italy (22):
  - Dipartimento Area Medica P.O., Ascoli Piceno
  - Unità Operativa Ematologica - Università degli Studi di Bari, Bari
  - Ospedali Riuniti, Bergamo
  - stituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Sezione di Ematologia e Trapianti Spedali Civili, Brescia
  - Azienda Spedali Civili, Brescia
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - Ospedale Ferrarotto, Catania
  - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro
  - Sezione di Ematologia e Fisiopatologia delle Emostasi - Azienda Ospedaliera - Arcispedale S. Anna, Ferrara
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Ospedale S. Luigi Gonzaga, Orbassano
  - La Maddalena Casa di Cura di Alta Specialità Dipartimento Oncologico di III Livello, Palermo
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - Ospedale S.Maria delle Croci, Ravenna
  - Calabria Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Università La Cattolica del Sacro Cuore, Roma
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - U.O. Ematologia, Azienda Ospedaliera Universitaria Senese, Siena
  - Policlinico Universitario - Clinica Ematologia, Udine
  - Policlinico G.B. Rossi, Verona

REFERENCES:
- [Background] Calabretta B, Perrotti D. The biology of CML blast crisis. Blood. 2004 Jun 1;103(11):4010-22. doi: 10.1182/blood-2003-12-4111. Epub 2004 Feb 24. PMID 14982876
- [Background] Barnes DJ, Melo JV. Management of chronic myeloid leukemia: targets for molecular therapy. Semin Hematol. 2003 Jan;40(1):34-49. doi: 10.1053/shem.2003.50002. PMID 12563610
- [Background] Goldman JM, Melo JV. Chronic myeloid leukemia--advances in biology and new approaches to treatment. N Engl J Med. 2003 Oct 9;349(15):1451-64. doi: 10.1056/NEJMra020777. No abstract available. PMID 14534339
- [Background] Goldman JM, Marin D, Olavarria E, Apperley JF. Clinical decisions for chronic myeloid leukemia in the imatinib era. Semin Hematol. 2003 Apr;40(2 Suppl 2):98-103; discussion 104-13. doi: 10.1053/shem.2003.50049. PMID 12783383
- [Background] Goldman JM, Marin D. Management decisions in chronic myeloid leukemia. Semin Hematol. 2003 Jan;40(1):97-103. doi: 10.1053/shem.2003.50009. PMID 12563616
- [Background] Goldman JM, Druker BJ. Chronic myeloid leukemia: current treatment options. Blood. 2001 Oct 1;98(7):2039-42. doi: 10.1182/blood.v98.7.2039. PMID 11567987
- [Background] Baccarani M, Russo D, Rosti G, Martinelli G. Interferon-alfa for chronic myeloid leukemia. Semin Hematol. 2003 Jan;40(1):22-33. doi: 10.1053/shem.2003.50004. PMID 12563609
- [Background] Martinelli G, Soverini S, Rosti G, Cilloni D, Baccarani M. New tyrosine kinase inhibitors in chronic myeloid leukemia. Haematologica. 2005 Apr;90(4):534-41. PMID 15820950
- [Background] Rosti G, Martinelli G, Bassi S, Amabile M, Trabacchi E, Giannini B, Cilloni D, Izzo B, De Vivo A, Testoni N, Cambrin GR, Bonifazi F, Soverini S, Luatti S, Gottardi E, Alberti D, Pane F, Salvatore F, Saglio G, Baccarani M; Study Committee, Italian Cooperative Study Group for Chronic Myeloid Leukemia; Writing Committee, Italian Cooperative Study Group for Chronic Myeloid Leukemia. Molecular response to imatinib in late chronic-phase chronic myeloid leukemia. Blood. 2004 Mar 15;103(6):2284-90. doi: 10.1182/blood-2003-07-2575. Epub 2003 Nov 26. PMID 14645009
- [Derived] Gugliotta G, Castagnetti F, Breccia M, Levato L, D'Adda M, Stagno F, Tiribelli M, Salvucci M, Fava C, Martino B, Cedrone M, Bocchia M, Trabacchi E, Cavazzini F, Usala E, Russo Rossi A, Bochicchio MT, Soverini S, Alimena G, Cavo M, Pane F, Martinelli G, Saglio G, Baccarani M, Rosti G; GIMEMA CML Working Party. Long-term outcome of a phase 2 trial with nilotinib 400 mg twice daily in first-line treatment of chronic myeloid leukemia. Haematologica. 2015 Sep;100(9):1146-50. doi: 10.3324/haematol.2015.129221. Epub 2015 Jun 25. PMID 26113419
- [Derived] Castagnetti F, Gugliotta G, Baccarani M, Breccia M, Specchia G, Levato L, Abruzzese E, Rossi G, Iurlo A, Martino B, Pregno P, Stagno F, Cuneo A, Bonifacio M, Gobbi M, Russo D, Gozzini A, Tiribelli M, de Vivo A, Alimena G, Cavo M, Martinelli G, Pane F, Saglio G, Rosti G; GIMEMA CML Working Party. Differences among young adults, adults and elderly chronic myeloid leukemia patients. Ann Oncol. 2015 Jan;26(1):185-192. doi: 10.1093/annonc/mdu490. Epub 2014 Oct 30. PMID 25361995
- [Derived] Lenaerts T, Castagnetti F, Traulsen A, Pacheco JM, Rosti G, Dingli D. Explaining the in vitro and in vivo differences in leukemia therapy. Cell Cycle. 2011 May 15;10(10):1540-4. doi: 10.4161/cc.10.10.15518. Epub 2011 May 15. PMID 21478667
- [Derived] Rosti G, Palandri F, Castagnetti F, Breccia M, Levato L, Gugliotta G, Capucci A, Cedrone M, Fava C, Intermesoli T, Cambrin GR, Stagno F, Tiribelli M, Amabile M, Luatti S, Poerio A, Soverini S, Testoni N, Martinelli G, Alimena G, Pane F, Saglio G, Baccarani M; GIMEMA CML Working Party. Nilotinib for the frontline treatment of Ph(+) chronic myeloid leukemia. Blood. 2009 Dec 3;114(24):4933-8. doi: 10.1182/blood-2009-07-232595. Epub 2009 Oct 12. PMID 19822896
- See also: GIMEMA's Web page — http://www.gimema.it